CLINICAL TRIAL: NCT05016648
Title: Cerebral Hemodynamics During Sustained Intra-operative Hypotension
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, D.P.Veelo, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: W20_244#20.270
Record Dates: First submitted 2021-08-17; First posted 2021-08-23 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Cerebral Autoregulation
Keywords: cerebral autoregulation; PEARS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PEARS patients: Patients who underwent the personalized external aortic root support procedure at the AMC. Cerebral monitoring measurements (NIRS, EEG, TCD and blood pressure) are used for the study.

SUMMARY:
Objective:

The objective of this study is to describe the physiology of the cerebral autoregulation over time during extreme low blood pressures (BP).

Study design:

This is a retrospective data collection study. During the Personalized External Aortic Root Support (PEARS) procedure extreme low blood pressures < 65 mmHg are medically induced. Hemodynamic and neurophysiologic data is for clinic purposes stored.

Study population:

All patients requiring a PEARS study at the Amsterdam University Medical Centers, location Amsterdam Medical Center (AMC).

Investigation:

Cerebral parameters during sustained low blood pressures are monitored with the transcranial doppler (TCD) for cerebral blood flow velocity (CBFV), near infrared spectroscopy (NIRS) for cerebral tissue oxygenation (rS02) and the electroencephalography (EEG) for the cerebral activity. Blood pressure waveforms are retrieved from an invasive arterial catheter. Besides, blood gasses during the low blood pressures and cardiac output, measured with a Schwan Ganz catheter are collected as well as electronic health records (EHR) (like age, gender and weight). All these devices are implemented as stated in the clinic protocol.

Main study parameters/endpoints:

The investigators will describe the cerebral autoregulation (CA) in several ways to retrieve a cut-off or lower limit of the CA where the regulation is either intact or impaired. First the static CA will be created with the mean arterial pressure (MAP) and mean cerebral blood flow (CBFm), second, the CA will be described with the mean flow velocity index (Mx, a method which calculates the correlation between the MAP and CBFm), COX (correlation between MAP and rS02) and with data of the EEG.

After retrieval of the cut off or lower limit, the CA below this point will be described over time to check for differences.

ELIGIBILITY:
Inclusion Criteria:

* Planned for a PEARS procedure
* Informed consent should be given

Exclusion Criteria:

* No informed consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients planned for the PEARS procedure at the AMC.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-08-07 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Cerebral autoregulation | During the entire operation, about 4 hours.
  A mechanism in the brain influenced by the cerebral blood pressure and cerebral blood flow velocity

CONTACTS AND LOCATIONS:
Locations (1):
- AUMC, Amsterdam, North Holland, Netherlands